CLINICAL TRIAL: NCT00302029
Title: Seroprevalence and Prospective Risk Factor Analysis of Cytomegalovirus (CMV) Infection in Adolescent Males
Brief Title: CMV Infection in Adolescent Males
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Director ORA, HHS/NIAID/DMID
Other Study IDs: 05-0126
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Cytomegalovirus Infections
Keywords: Cytomegalovirus, risk factors, seroprevalence
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and salvia samples.

GROUPS / COHORTS (2):
- CMV positive: CMV +, N=500/167
- CMV negative: CMV -, N=500/167

SUMMARY:
The purpose of this study is to find out more about cytomegalovirus (CMV) and how it is spread between people. One thousand adolescent males ages 12-17 years will participate in this study. Participants will be given a questionnaire about risk factors for CMV. A small blood sample (2-3 teaspoons) will be taken to test for CMV infection. Subjects that are CMV seronegative may participate in the second part of this study, which will involve returning to the clinic at regularly scheduled visit times to provide blood, urine, and saliva (spit) samples. This part of the study will take at least 24 months to complete. Subjects that test positive for CMV during the 2nd portion of the study will be invited to participate in the 3rd part of the study. This part of the study will require 8 regularly scheduled visits to provide blood, urine and saliva samples, over a 12-month period. The maximum amount of time a subject will participate in the study is 36 months.

DETAILED DESCRIPTION:
The objectives of this study are to: (1) to determine the prevalence of cytomegalovirus (CMV) infection and risk factors for infection in adolescent males; (2) to prospectively define the incidence and to evaluate risk factors for acquisition of CMV infection in adolescent males; and (3) to provide preliminary data on the duration and magnitude of CMV in the urine, saliva, and blood in those subjects who seroconvert during the study. Approximately 1000 males aged 12 to 17 years will be recruited from adolescent clinics at Cincinnati Children's Hospital Medical Center, Vanderbilt University, and the University of Texas Medical Branch at Galveston in order to obtain 225 CMV-seronegative subjects (75 at each site) to complete the Prospective Risk Factor Analysis. Patient participation will last a minimum of 24 months with 8 scheduled visits for the prospective seroepidemiology study. Patients who seroconvert will be invited to join the viral load analysis portion of the study, which consists of 8 scheduled visits during a 12 month period. The maximum duration of the study is 36 months, but will depend on the timing of seroconversion and entry into the viral load analysis. The study is divided into 3 parts: Seroprevalence, Prospective Risk Factor Analysis, and Prospective Viral Load Analysis. In the Seroprevalence portion of the study, after subjects have completed informed assent and parents or guardian consent, a small amount (10 mL) of blood will be obtained from subjects for evaluation of CMV antibody by commercial ELISA. Participants will be given a CMV fact sheet. Subjects will be contacted by phone with results of CMV antibody testing and the implications. They will be given the opportunity to receive the fact sheet again and discuss this information with study personnel, if they desire. Also at this visit, subjects who meet the eligibility criteria will be asked to complete a detailed questionnaire regarding possible risk factors for CMV infection. For those subjects 14 years of age and older, the questionnaire will include questions about sexual practices. Risk factors for CMV infection will then be compared between those subjects who are seropositive and those who are seronegative. Subjects who are CMV seronegative will be invited to participate in the Prospective Risk Factor Analysis portion of the study to determine the incidence of CMV infection and risk factors for acquisition in adolescent males. Eligible subjects will be identified and provided with a description of the study by a research nurse or study coordinator. Subjects will be asked to sign a separate assent and consent will be obtained from the parent or legal guardian. It is anticipated that recruitment will require approximately 1 year. Every 3 months, urine (For CMV culture and polymerase chain reactions [PCR]) and serum samples (for CMV antibody and PCR) will be collected from the subjects and analyzed for identification of CMV infection. In addition, subjects will complete a questionnaire evaluating risk factors at each 3-month visit. For those subjects who are 14 years of age or older, the questionnaire will include questions about sexual practices. If the subject tests positive for CMV, he will be asked to sign a separate consent to participate in the third phase of the study. In the Prospective Viral Load Analysis, subjects who seroconvert during the second portion of the study will be invited to participate in an evaluation of the duration and magnitude of CMV levels in blood, urine, and saliva. Subjects will be seen every month for 4 months followed by every 2 months for 8 months for collection of these specimens.

ELIGIBILITY:
Inclusion Criteria: 1. Subjects must be willing and able to provide written informed assent prior to enrollment, and parent(s) or legal guardian must provide written informed consent prior to study enrollment. 2. Subjects must be male and between 12 to 17 years of age at the time of initial study entry. 3. Subjects must be willing and able to comply with the requirements of the protocol and must be available for the 24-month duration of the study (for Prospective Risk Factor Analysis portion of the study only). 4. Subjects must be willing and able to comply with the requirements of the protocol and must be available for the 12-month duration of the study (for CMV Viral Load Analysis). Exclusion Criteria: 1. Receipt of blood and/or blood products in the past 3 months (Subjects meeting this exclusion criterion will also be excluded from the Seroprevalence study visit); 2. Unable to comply with the study protocol; 3. Infection with CMV prior to Seroprevalence study (for Prospective Risk Factor Analysis and CMV Viral Load Analysis portions of the study only); 4. History of any physical, mental or developmental disorder that study personnel believe may hinder a participant's ability to comply with study requirements (for Prospective Risk Factor Analysis and CMV Viral Load Analysis portions of the study only); 5. History of malignancy or having a confirmed or suspected immunodeficient condition such as HIV infection or receipt of immunosuppressive drugs. Inhaled and topical corticosteroids will be allowed (for Prospective Risk Factor Analysis and CMV Viral Load Analysis portions of the study only); 6. Receipt of or history of receipt of any medications or treatments that affect the immune system, such as immune globulin, interferon, immunomodulators, cytotoxic drugs, or other drugs known to be frequently associated with significant major organ toxicity or systemic steroids (oral or injectable) in the past 6 months (for Prospective Risk Factor Analysis and CMV Viral Load Analysis portions of the study only); 7. Prior receipt of a CMV vaccine.

Ages: 12 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1000 males aged 12 - 17 years will be recruited from participating adolescent clinics at Cincinnati Children's Hospital Medical Center (CCHMC), Vanderbilt University Medical Center, and the University of Texas Medical Branch Galveston.
Sampling Method: Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of CMV infection in adolescent boys | Obtained every month for 4 months and then every 2 months for 8 months.
Prospectively determine the incidence of CMV infection. | Day 0 and every 3 months for 24 months.
Determine the duration and magnitude of CMV replication in the blood, urine, and saliva by specimens. | Obtained every month for 4 months and then every 2 months for 8 months.

SECONDARY OUTCOMES:
Prospectively identify risk factors for infection. | Day 0 and every 3 months for 24 months.
Identify risk factors for CMV infection by comparing those subjects who are CMV seropositive with those subjects who are CMV seronegative. | Screening

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - The University of Texas Medical Branch, Galveston, Texas